CLINICAL TRIAL: NCT05099094
Title: A Safety and Efficacy Study of VEGFA-targeting Gene Therapy to Treat Refractory Retinal and Choroidal Neovascularization Diseases
Brief Title: VEGFA-targeting Gene Therapy to Treat Retinal and Choroidal Neovascularization Diseases
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai BDgene Co., Ltd. (Industry)
Collaborators: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BD311
Record Dates: First submitted 2021-09-18; First posted 2021-10-29 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2024-06

CONDITIONS: Neovascular Age-related Macular Degeneration; Diabetic Macular Edema; Retinal Vein Occlusion
Keywords: Retinal diseases; Choroidal diseases; Neovascularization; nAMD; neovascular age-related macular degeneration; DME; Diabetic macular edema; RVO-ME; Retinal vein occlusion-Macular edema
MeSH Terms: conditions — Retinal Vein Occlusion; Retinal Diseases; Choroid Diseases; Neovascularization, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BD311 Adults single group (Experimental): Administered by suprachoroidal injection. Dosage form: injection solution. Dose: 500uL. Frequency of administration: one time injection.
  Interventions: Genetic: BD311

INTERVENTIONS:
Genetic: BD311 — Integration-deficient lentiviral vector (IDLV) expressing VEGFA antibody

SUMMARY:
Patients who respond to anti-VEGF therapy but with refractory retinal and choroidal neovascularization diseases including neovascular age-related macular degeneration (nAMD), diabetic macular edema (DME), and retinal vein occlusion-Macular edema (RVO-ME).

DETAILED DESCRIPTION:
Choroidal and retinal angiogenesis diseases are a group of diseases characterized by choroidal or retinal angiogenesis. These diseases are often correlated with the macular area, which may lead to significant visual loss. In this study, The IDLV vector is engineered to carry the VEGFA antibody gene. The gene is delivered to the RPE cells to express the VEGFA antibody which neutralizes the VEGFA activity in the posterior segment of the eye of individuals who have progressed to various forms of neovascular macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with nAMD at the age ≥50; Or patients with diabetic macular edema (DME) at the age ≥18; Or patients with macular edema following retinal vein occlusion (RVO-ME) at the age ≥18.
2. Early Treatment Diabetic Retinopathy Study (ETDRS) best corrected visual acuity ≤63 and letter score ≥19 Corresponding Snellen vision ≤20/63 and ≥20/400).
3. OCT confirms the presence of intraretinal fluid or subretinal fluid in the fovea.
4. Have received anti-VEGF therapy in the past and have responded to anti-VEGF therapy.
5. With refractory conditions: repeated anti-VEGF treatments are required due to the disease condition. When the treatment is interrupted, the disease condition recurs (OCT examination indicates increased subretinal/inner effusion in the macula)
6. For patients with both eyes suffered, enroll the one with more severe condition.
7. Routine blood test, liver and kidney function, coagulation index of patients is normal：AST/ALT < 2.5 × ULN; TB < 1.5 × ULN; PT < 1.5 × ULN; Hb > 10 g/dL (male) and > 9 g/dL (female); PLT > 100 × 10^3/µL; eGFR > 30 mL/min/1.73 m^2.

Subjects voluntarily join the study, sign an informed consent form, have good compliance, and cooperate with follow-up.

Exclusion Criteria:

1. Choroidal neovascularization or macular edema induced by other diseases.
2. Any other factors that affect vision improvement in the study eye, such as fibrosis, atrophy, or RPE tear in the fovea of the macula.
3. The study eye already has severe proliferative retinopathy, such as retinal neovascularization, traction retinal detachment, etc. (only for DME and RVO-ME patients) .
4. Retinal detachment or advanced glaucoma in the study eye.
5. Implants in the study eye (except intraocular lenses).
6. Received internal eye surgery within 3 months prior to enrollment.
7. Vitrectomy surgery on the study eye.
8. Received intravitreal glucocorticoid or other clinical research drugs (except anti-VEGF therapy) within 6 months prior to enrollment.
9. Myocardial infarction, cerebrovascular accident or transient ischemic attack occurred within 6 months prior to enrollment.
10. Poorly controlled hypertension under maximum medication (systolic blood pressure>180 mmHg, diastolic blood pressure>100 mmHg).
11. Poor blood glucose control under medication (fasting blood glucose is greater than or equal to 10.0 umol/L).
12. Women who are willing to give birth; pregnant/breastfeeding women Have received gene therapy in the past.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Treatment-related adverse events | At multiple timepoints after infusion up to 12 months.
  Observe and record incidences of AE and SAE related to VEGFA-targeting gene therapy drug BD311 (IDLV expressing VEGFA antibody) administration.

SECONDARY OUTCOMES:
Changes in macular intraretinal fluid (IRF) | At multiple timepoints after infusion up to 12 months.
  The presence of macular intraretinal fluid (IRF) will be determined by optical coherence tomography (OCT).
Changes in subretinal fluid (SRF) | At multiple timepoints after infusion up to 12 months.
  The presence of subretinal fluid (SRF) will be determined by optical coherence tomography (OCT).
Change in central retinal thickness (CRT) | At multiple timepoints after infusion up to 12 months.
  Central retinal thickness will be measured by Optical Coherence Tomography (OCT).
Changes in the area of choroidal neovascularization | At multiple timepoints after infusion up to 12 months.
  Using Fluorescein angiography (FFA) and indocyanine green angiography (ICGA) to assess the areas of choroidal neovascularization. Only for patients with nAMD.
Changes in the area of fluorescein leakage | At multiple timepoints after infusion up to 12 months.
  Using Fluorescein angiography (FFA) and indocyanine green angiography (ICGA) to assess the areas of fluorescein leakage. Only for patients with nAMD.
The number of rescue treatments | At multiple timepoints after infusion up to 12 months.
  Rescue treatments that require vitreous anti-VEGF injections due to illness.
Evaluate the visual improvement | At multiple timepoints after infusion up to 12 months.
  Subjects will be examined for best corrected visual acuity (BCVA).

CONTACTS AND LOCATIONS:
Overall Officials: Gezhi Xu, Dr, Study Director — Eye & ENT Hospital of Fudan University
Locations (1):
- Eye & ENT Hospital of Fudan University, Shanghai, SH, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Romano F, Lamanna F, Gabrielle PH, Teo KYC, Battaglia Parodi M, Iacono P, Fraser-Bell S, Cornish EE, Nassisi M, Viola F, Agarwal A, Samanta A, Chhablani J, Staurenghi G, Invernizzi A. Update on Retinal Vein Occlusion. Asia Pac J Ophthalmol (Phila). 2023 Mar-Apr 01;12(2):196-210. doi: 10.1097/APO.0000000000000598. Epub 2023 Feb 14. PMID 36912792